CLINICAL TRIAL: NCT04542083
Title: Impact of COVID-19 on Unplanned Admissions for Acute Cardiovascular and Neurovascular Conditions in France
Brief Title: Covid-19, Acute Myocardial Infarctions and Strokes in France
Acronym: COVUSI
Status: Terminated | Type: Observational
Why Stopped: Maximum recruitment reached
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0513
Record Dates: First submitted 2020-09-04; First posted 2020-09-09 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Acute Cardiovascular Condition; Acute Neurovascular Condition; Stroke; Acute Myocardial Infarction
MeSH Terms: conditions — COVID-19; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 period: Admissions from January to December 2020
- Control period: Admissions from January 2018 to December 2019

SUMMARY:
The COVID-19 pandemic has had dramatic effects on health systems and on non-COVID health care.

Using French inpatient claims data and retrospectively collected clinical data, the investigators will assess the changes in hospital admissions for acute cardiovascular and neurovascular conditions in France during and after the national lockdown.

ELIGIBILITY:
Inclusion criteria:

- Adults admitted in 2018, 2019 or 2020 in a French hospital for acute coronary syndrom or stroke

Exclusion criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Daily number of admissions for acute cardio- and neurivascular conditions in France. | 1 day
  Daily number of admissions for acute cardio- and neurivascular conditions in France.

SECONDARY OUTCOMES:
Specific mortality rate. | 1 day
  Specific mortality rate.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Mercier, PU PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC